CLINICAL TRIAL: NCT03276208
Title: Pregnancy Massage and Mindfulness Study for Tobacco Smoking Women
Brief Title: Pregnancy, Mindfulness, and Massage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of enrollment.
Sponsor: Yale University (Other)
Collaborators: Massage Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000021692
Record Dates: First submitted 2017-08-20; First posted 2017-09-08 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Tobacco Use; Pregnancy Related
Keywords: Pregnancy; Tobacco; Massage Therapy; Mindfulness
MeSH Terms: conditions — Tobacco Use | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Masking Description: During initial telephone screening participants will be randomized to either intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Therapy and Mindfulness (Experimental): Participants in the intervention group will receive two prenatal massages a week for a three-week period. They will also be enrolled in the mindfulness-based Craving to Quit® tobacco cessation program during this 3-week period.
  Interventions: Other: Prenatal Massage; Other: Mindfulness
- Mindfulness (Active Comparator): Participants will enroll in the mindfulness-based Craving to Quit® tobacco cessation program during the same 3-week period. A massage will be provided upon completion of the study.
  Interventions: Other: Mindfulness

INTERVENTIONS:
Other: Prenatal Massage — We will utilize moderate pressure Swedish massage (SM) that utilizes long slow strokes known as effleurage and kneading strokes known as petrissage. A specific routine will be performed on each participant with focus on low back, upper back, shoulders, and neck musculature. Consistent moderate pressure, which is lighter than deep tissue massage but deeper than brush strokes, will be used.
  Arms: Massage Therapy and Mindfulness
Other: Mindfulness — The intervention and control group will be enrolled in the Craving to Quit® program, a 21-day mindfulness-based program delivered via a smartphone application (https://www.cravingtoquit.com/). This program uses a mindfulness-based approach to train people to recognize and be aware of their tobacco cravings. The program includes videos, online exercises to complete, and a virtual support community.

SUMMARY:
This trial will examine the contribution of massage therapy and mindfulness to tobacco-smoking women in the third trimester of pregnancy.

DETAILED DESCRIPTION:
Massage therapy may be a viable approach to decrease stress during pregnancy that may in turn reduce tobacco consumption. Massage therapy may not be sufficient as a stand-alone approach, and may be better suited partnered with a cessation approach that targets another mechanism of addiction, craving. Therefore, participants (N=60) will be enrolled in the Craving to Quit® tobacco cessation program, designed by researchers at Yale, which employs a mindfulness-based approach to train participants to recognize and bring cravings into their conscious awareness. Each mother will be randomly assigned to a bi-weekly massage intervention (n=30) or control (n=30) group. Participants in the intervention group will receive two prenatal massages a week for a three-week period.

ELIGIBILITY:
Inclusion Criteria:

* currently pregnant in third trimester
* singleton pregnancy
* aged 18 years or older
* women smoked before their pregnancy
* women who currently smoke at least 5 cigarettes per day at enrollment
* women need access to a smartphone
* women expressing an interest in learning skills to help decrease tobacco-smoking

Exclusion Criteria:

* incapable of giving informed consent
* insufficient English fluency
* participating in other smoking cessation programs
* evidencing severe psychiatric symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on biological sex as study of pregnancy
Enrollment: 12 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Tobacco Use Change from Baseline to Post-Intervention | Up to 4 weeks
  Number of cigarettes smoked in past 24 hours
Withdrawal Symptoms Change from Baseline to Post-Intervention | Up to 4 weeks
  Mood and Physical Symptoms Scale
Nicotine Dependence Change from Baseline to Post-Intervention | Up to 4 weeks
  FTND (Fagerstrom Test for Nicotine Dependence) measure
Depression Change from Baseline to Post-Intervention | Up to 4 weeks
  EPDS (Edinburgh Postnatal Depression Scale) measure
Anxiety Change from Baseline to Post-Intervention | Up to 4 weeks
  Beck Anxiety Inventory
Stress Change from Baseline to Post-Intervention | Up to 4 weeks
  Perceived Stress Scale
Daily Stress Scores Change from Baseline to Post-Intervention | Up to 4 weeks
  Diary Measure
Daily Tobacco Usage Change from Baseline to Post-Intervention | Up to 4 weeks
  Diary Measure
Heart Rate Variability Change from Baseline to Post-Intervention | Up to 4 weeks
  Maternal heart rate variability measured at rest

SECONDARY OUTCOMES:
Neonatal Outcomes | Up to 2 months
  mode of delivery (including any complications), infant well-being, gestational age, and weight.
Fetal Heart Rate Change from Baseline to Post-Intervention | Up to 4 weeks
  Fetal heart rate measured at rest
Engagement with Craving to Quit | Up to 4 weeks
  Engagement with the Craving to Quit app

OTHER OUTCOMES:
CO (carbon monoxide) monitoring Change from Baseline to Post-Intervention | Up to 4 weeks
  breath test
MINI (Mini International Neuropsychiatric Interview) Substance Dependence | Enrollment
  determine other substance use disorders
Self-Reported Mood at each Massage Therapy Session for Intervention Group | Up to 3 weeks
  positive and negative mood, including stress
Mind-mindedness related to infant | Up to 2 months
  Describe your child measure; this will be a narrative statement provided by participants where they are asked to describe their child. These narratives will be scored to ascertain the total number of mind-minded comments included in the narrative.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Rutherford, PhD, Principal Investigator — Yale University; Michael Paidas, MD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No